CLINICAL TRIAL: NCT05524519
Title: Intradermal Acupuncture Based on Changes in Biological Specificity of Acupoints for Major Depressive Disorder: a Prospective, Multicentre, Randomized, Controlled Trial
Brief Title: Intradermal Acupuncture Based on Changes in Biological Specificity of Acupoints for Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Collaborators: Zhejiang Provincial Tongde Hospital (Other); First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Xiaomei Shao, Prof, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022ZX010-BIA
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Intradermal acupuncture; Biological specificity
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Dosage Forms; theasinensin A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- WL group (Active Comparator): This group will include 40 patients with MDD. Patients in this group will not receive IA treatment during the study period. When the study is over, they will receive 6 weeks of the same IA treatment as in the CCA group.
  Interventions: Drug: Basic treatment
- CCA group (Experimental): This group will include 40 patients with MDD who will be treated with basic treatment and IA. LR3, PC6, SP6, and HT7 will be selected for IA.
  Interventions: Drug: Basic treatment; Procedure: CCA
- TSA group (Experimental): This group will include 40 patients with MDD who will be treated with basic treatment and IA. TSA selected in the first part of the study will be stimulated.
  Interventions: Drug: Basic treatment; Procedure: TSA
- PSA group (Experimental): This group will include 40 patients with MDD who will be treated with basic treatment and IA. PSA selected in the first part of the study will be stimulated.
  Interventions: Drug: Basic treatment; Procedure: PSA

INTERVENTIONS:
Drug: Basic treatment — 1. Health education: Properly explain the causes and precautions of the patient and instruct the patient to rest regularly. In addition, care should be enhanced to avoid accidents.
  2. The basic therapeutic drug is the use of one or more antidepressants, such as oral 5-hydroxytryptamine reuptake inhibitors, dual inhibitors of pentraxin and norepinephrine reuptake, noradrenergic and specific pentraxinergic antidepressants, pentraxin receptor balance antagonists, tricyclic antidepressants, etc. If there is significant sleep disturbance, benzodiazepines may be added temporarily. Dosing and dosage will be adjusted by a specialist.
  Other Names: Health education and medication
Procedure: PSA — Four PSA selected in the first part of the study will be stimulated. According to the position of the acupoints, choose a needle of φ0.20*1.5m or φ0.20*1.2mm. Press the needle to insert the acupoint vertically and retain it in the skin. After the intervention, the needle will be retained for 72 hours with a day of rest after removal. During needle retention, participants will be instructed to press the acupoints 3-4 times a day for about 1 minute each time, with the amount of stimulation as much as the patient can tolerate, at an interval of about 4 hours. A total of 10 treatment sessions will be performed for 6 weeks.
  Other Names: Intradermal acupuncture in PSA
  Arms: PSA group
Procedure: TSA — Four TSA selected in the first part of the study will be stimulated. According to the position of the acupoints, choose a needle of φ0.20*1.5m or φ0.20*1.2mm. Press the needle to insert the acupoint vertically and retain it in the skin. After the intervention, the needle will be retained for 72 hours with a day of rest after removal. During needle retention, participants will be instructed to press the acupoints 3-4 times a day for about 1 minute each time, with the amount of stimulation as much as the patient can tolerate, at an interval of about 4 hours. A total of 10 treatment sessions will be performed for 6 weeks.
  Other Names: Intradermal acupuncture in TSA
  Arms: TSA group
Procedure: CCA — Acupoints: LR3 (Taichong), PC6 (Neiguan), SP6 (Sanyinjiao), and HT7 (Shengmen). PC6 and HT7 will use φ0.20*1.2mm acupuncture needle. LR3 and SP6 will use φ0.20*1.5m acupuncture needles. Press the needle to insert the acupoint vertically and retain it in the skin. After the intervention, the needle will be retained for 72 hours with a day of rest after removal. During needle retention, participants will be instructed to press the acupoints 3-4 times a day for about 1 minute each time, with the amount of stimulation as much as the patient can tolerate, at an interval of about 4 hours. A total of 10 treatment sessions will be performed for 6 weeks.
  Other Names: Intradermal acupuncture in CCA
  Arms: CCA group

SUMMARY:
Acupoints are the stimulus points and reactive points for acupuncture to treat diseases. Therefore, this study is designed to detect the pain threshold and temperature of biological specificities of acupoints in healthy control (HC) participants and major depressive disorder (MDD) participants by using pressure pain threshold gauge (PTG) and infrared thermography (IRT). Based on the results of the PTG and IRT tests, the potentially superior acupoints for the treatment of MDD will be selected separately. Then, different acupoint groups selected based on different biological specificities tests will be used for clinical treatment to evaluate the clinical efficacy of intradermal acupuncture (IA) for MDD based on changes in the biological specificities of acupoints.

DETAILED DESCRIPTION:
Part 1: This study will include 50 patients with MDD (MDD group) and 50 HC participants (HC group). PTG and IRT, respectively, will be adopted to assess 2 kinds of biological specificity of MDD-related acupoints: pain sensitivity specificity and thermal specificity. Based on the results of the PTG and IRT tests, the potentially superior acupoints for the treatment of MDD will be selected separately. After statistical analysis of the data from PTG and IRT tests, 4 pressure pain threshold strong response acupoints (PSA) and 4 temperature strong response acupoints (TSA) will be selected, respectively. This part of the trial began on January 10, 2022, and its registration number is NCT06114342.

Part 2: A total of 160 participants with MDD who meet the inclusion criteria will be included in the study. Patients with MDD who met the criteria will be randomly divided 1:1:1:1 into 4 groups: wait-listed treatment (WL) group, clinical common acupoint (CCA) group, TSA group, and PSA group. All participants received basic therapeutic medication for the use of one or more antidepressants. Dosing and dosage will be adjusted by a specialist. The Patient Health Questionnaire-9 (PHQ-9) and the MOS item short form health survey (SF-36) will be used as clinical efficacy outcome indicators, and each group's incidence of adverse effects will be observed. This study will investigate the effectiveness and safety of IA based on changes in the biological specificity of acupoints for MDD.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for HC:

* HC who could provide a recent depression screening report, and confirm they have not any cardiovascular, respiratory, digestive, urinary, hematological, endocrine, or neurological disease;
* 18 ≤ age ≤60 years, male or female;
* Participants have clear consciousness and could communicate with others normally;
* Participants could understand the full study protocol and have high adherence. Written informed consent is signed by themselves.

Inclusion criteria for MDD:

* Patients should meet the diagnostic criteria of the International Classification of Diseases 10th Edition (ICD-10) diagnostic criteria for MDD;
* 18 ≤ age ≤60, male or female;
* Participants have clear consciousness and could communicate with others normally;
* Participants could understand the full study protocol and have high adherence. Written informed consent is signed by themselves.

Exclusion Criteria:

Exclusion criteria of HC:

* Participants with serious primary diseases of cardiovascular diseases, liver diseases, kidney diseases, urinary diseases, and hematological diseases;
* Participants have a mental illness, alcohol dependence, or a history of drug abuse;
* Pregnant or lactating participants;
* Participants with intellectual disabilities who cannot cooperate with the questionnaire survey;
* Participants with bleeding tendency, skin disease, allergic constitution, and allergic to adhesive tape;
* The skin at the test site of participants has scars, hyperpigmentation, red and swollen;
* Participants are participating in other trials.

Exclusion criteria for MDD:

* Participants with serious primary diseases of cardiovascular, respiratory, digestive, urinary, hematological, endocrine, neurological disease, and other serious primary diseases, and the disease cannot be effectively controlled clinically;
* MDD caused by organic mental disorders, schizophrenia, bipolar disorder, psychoactive substances, and non-addictive substances;
* Participants with suicidal tendencies;
* Pregnant or lactating participants;
* Participants with intellectual disabilities who cannot cooperate with the questionnaire survey;
* Participants with bleeding tendency, skin disease, allergic constitution, and allergic to adhesive tape;
* The skin at the test site of participants has scars, hyperpigmentation, red and swollen. IRT is not be performed on female subjects during their menstrual and ovulatory periods;
* Participants are participating in other trials.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the Patient Health Questionaire-9 Items (PHQ -9) | Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up.
  The PHQ-9 scale has a total of 9 questions, each with a score of 0-3 (none: 0; a few days: 1; more than half of the time: 2; almost every day: 3), with a total score of 0-27.

SECONDARY OUTCOMES:
Change in the MOS item short form health survey (SF-36) | Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up.
  The SF-36 scale evaluates the quality of healthy life into 8 dimensions, which are divided into two categories: physical health and mental health, namely physical function (PF), role physical (RP), body pain (BP), general health (GH), vitality (VT), social function (SF), role emotional (RE), mental health (MH).
Temperature change of relevant sites | Baseline, 6 weeks after treatment.
  NEC R450 Infrared thermography will be used to record baseline temperature and the temperature change of relevant sites. The average temperature value of relevant sites in the six infrared thermograms is its base temperature.
Pain sensitivity change of relevant sites | Baseline, 6 weeks after treatment.
  A pressure pain threshold gauge will be used to measure the local pain threshold (PT). The probe of the pain gauge will be placed vertically on the relevant test site, and the pressure will be applied slowly and steadily, and when the participant feels pain, the pressure will stop and the reading on the gauge is the PT. The average value of the PT of the same relevant test sites will be calculated as their base PT.
Adverse Events | through study completion (up to 10 weeks).
  The adverse events that occurred during the study will be recorded, including symptoms, signs, the time of appearance, duration, degree of severity, treatment measures, and the course of treatment, and their correlation with the treatment will be evaluated.
  Incidence of adverse events = number of cases of adverse events /total number of cases in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Shao, Ph.D, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tu M, Wu X, Qu S, Jin J, Chen N, Xiong S, Pei S, Li X, Shi Y, Hu H, Li X, Fang J, Shao X. The effective on intradermal acupuncture based on changes in biological specificity of acupoints for major depressive disorder: study protocol of a prospective, multicenter, randomized, controlled trial. Front Psychiatry. 2023 Jun 9;14:1183127. doi: 10.3389/fpsyt.2023.1183127. eCollection 2023. PMID 37441145